CLINICAL TRIAL: NCT01495520
Title: Ranolazine for the Treatment of sYmPtoms of PaLpitations in patiEnts With Ischemic Heart Disease - The RYPPLE Trial
Brief Title: Ranolazine for Improving Symptoms of Palpitations
Acronym: RYPPLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 671/2011/D
Record Dates: First submitted 2011-12-15; First posted 2011-12-20 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Ischemic Heart Disease
Keywords: Arrhythmias; palpitations
MeSH Terms: conditions — Myocardial Ischemia; Arrhythmias, Cardiac | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Patients will receive ranolazine 750 mg bid for 30 days
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Patients will receive placebo for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — os, pill, 750 mg, b.i.d., 30 days
  Other Names: Ranexa TM, Gilead, US
  Arms: Ranolazine
Drug: Placebo — os, pill, b.i.d., 30 days
  Arms: Placebo

SUMMARY:
Patients with ischemic heart disease often report multiple symptoms, including angina and palpitations. Ranolazine has antiarrhythmic effects which are largely a result of the drug's effect on multiple ion channels. It remains unknown, however, whether the favorable effects of ranolazine on symptoms and arrhythmias are maintained over time. Aim of this study is to test the hypothesis that chronic treatment with ranolazine can improve the symptomatic status of patients with ischemic heart disease by reducing the occurrence of palpitations.

DETAILED DESCRIPTION:
Background:

Patients with ischemic heart disease often report multiple symptoms, including angina and palpitations.

Ranolazine is a novel antianginal and antiischemic drug that reduces intracellular sodium and calcium accumulation during ischemia thus limiting ischemic injury. Furthermore, ranolazine has antiarrhythmic effects which are largely a result of the drug's effect on multiple ion channels.

It has previously been shown that treatment with ranolazine can reduce the frequency of supraventricular and ventricular tachycardia in the short term. In a subgroup analysis of the MERLIN-TIMI 36 trial, the continuous ECGs of 6,351 patients were analyzed. The results showed that, in comparison with placebo, treatment with ranolazine resulted in fewer episodes of ventricular tachycardia that lasted 8 beats or longer (5.3% versus 8.3%; P <0.001), and in fewer episodes of supraventricular tachycardia (44.7% versus 55%; P <0.001) and new-onset atrial fibrillation (1.7% versus 2.4%; P=0.08).

It remains unknown, however, whether the favorable effects of ranolazine on symptoms and arrhythmias are maintained over time.

Purpose:

The primary objective of this study is to test the hypothesis that chronic treatment with ranolazine can improve the symptomatic status of patients with ischemic heart disease by reducing the occurrence of palpitations.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of palpitations
* Angiographically-proven coronary artery disease
* Stable conditions
* No recent acute coronary syndromes
* Able to understand and willing to sign the informed consent form
* Symptomatic patients (palpitation) with stable angina pectoris already on therapy with beta-blockers and/or calcium antagonists.

Exclusion Criteria:

* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours
* Severe renal failure
* Severe hepatic failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of symptoms of palpitations | Up to 30 days
  Occurrence of symptoms of palpitations

SECONDARY OUTCOMES:
Occurrence of arrhythmia in case of symptoms of palpitations | Up to 30 days
  Definition of presence, number, type and duration of the arrhythmia in case of the patient-reported symptoms of palpitations

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University Sapienza